Official Title: AN OPEN-LABEL STUDY OF THE LONG-TERM SAFETY AND TOLERABILITY OF SAGE-324 IN PARTICIPANTS WITH ESSENTIAL TREMOR

NCT ID: NCT05366751

Document Date: Statistical Analysis Plan Version 1.0 23 October 2024

# 9. STATISTICAL METHODS INTERIM ANALYSIS PLAN

The following statistical analysis plan is provided:

Sage\_324-ETD-303\_sap\_v10\_20241022



# STATISTICAL ANALYSIS PLAN METHODS PROTOCOL NUMBER 324-ETD-303

An Open-label Study of the Long-term Safety and Tolerability of SAGE-324 in Participants with Essential Tremor

Author(s) of SAP:

:

Version: 1.0

Version Date of SAP: 22 October 2024

Sponsor:

Sage Therapeutics, Inc. 55 Cambridge Parkway Cambridge, Massachusetts 02142

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Sage Therapeutics, Inc. is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

Sage Therapeutics, Inc. CONFIDENTIAL

## Authorization Signature Page

An Open-label Study of the Long-term Safety and Tolerability of SAGE-324 in Participants with Essential Tremor



| Statistical Analysis Plan Methods Version 1.0 22Oct2024 | Sage Therapeutics, Inc. |
|---|---|
| Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) | CONFIDENTIAL |
| | 22 0-4 2024 11.50 502 |
| | 23-Oct-2024 11:50 ED1 |
| PhD | Date |

Sage Therapeutics, Inc

Sage Therapeutics, Inc. CONFIDENTIAL

# TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS | 6 |
|--------|-----------------------------------------------------------|----|
| 2. | INTRODUCTION | 7 |
| 3. | STUDY OBJECTIVES | 8 |
| 3.1. | Primary Objective | 8 |
| 3.2. | Secondary Objective | 8 |
| | | 8 |
| 4. | STUDY ENDPOINTS | 9 |
| 4.1. | Primary Endpoint | 9 |
| 4.2. | Secondary Endpoints | 9 |
| | | 9 |
| 5. | STUDY DESIGN | 10 |
| 5.1. | Overall Design | 10 |
| 5.2. | Sample Size and Power | 11 |
| 5.3. | Randomization | 11 |
| 5.4. | Blinding and Unblinding | 11 |
| 6. | MODIFICATIONS | 12 |
| 6.1. | Modifications from the Approved Clinical Study Protocol | 12 |
| 6.2. | Modifications from the Approved Statistical Analysis Plan | 12 |
| 6.3. | Modifications from the Approved DMC Charter | 12 |
| 7. | ANALYSIS SETS | 13 |
| 7.1. | All Participants Set | 13 |
| 7.2. | Safety Set | 13 |
| | | 13 |
| | | 13 |
| 8. | STATISTICAL ANALYSIS | 14 |
| 8.1. | General Considerations | 14 |
| 8.2. | Background Characteristics | 14 |
| 8.2.1. | Participant Disposition. | 14 |
| 8.2.2. | Protocol Deviations | 15 |
| 8.2.3. | Demographics and Baseline Characteristics | 15 |

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL 8.2.4. 8.2.5. Prior and Concomitant Medications \_\_\_\_\_\_\_\_16 8.2.6. 8.2.7. 18 18 18 19 19 21 8.4 8.4.1. Adverse Events 23 8.4.2. Clinical Laboratory 24 8.4.3. Electrocardiogram 27 8.4.4. 8.4.5. 8.4.6. 8.4.7. 8.4.8. 8.4.9. 8.6. 9 9.1. 9.2. REFERENCES 33 10. 11. 

Sage Therapeutics, Inc. CONFIDENTIAL

# 1. LIST OF ABBREVIATIONS

The following abbreviations and specialist terms are used in this statistical analysis plan (SAP).

Table 1: Abbreviations and Specialist Terms

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AE | adverse event |
| BMI | body mass index |
| COVID-19 | Coronavirus disease 2019 |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOS | End of Study |
| EOT | End of Treatment |
| ESS | Epworth Sleepiness Scale |
| ET | essential tremor |
| IP | investigational product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PWC-20 | 20-item Physician Withdrawal Checklist |
| QTcF | QT corrected according to Fridericia's formula |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | System Organ Class |
| TEAE | treatment-emergent adverse event |
| WHO-DD | World Health Organization Drug Dictionary |

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

## 2. INTRODUCTION

This statistical analysis plan (SAP) is for the final analysis of Study 324-ETD-303 and is based on the approved clinical study protocol dated 02 Nov 2023, Version 4.0.

This SAP addresses the objectives of the study and describes the planned statistical analyses and data presentations. All analyses and data presentations will be generated using SAS® Version 9.4 or higher software (SAS Institute, Cary, North Carolina, USA). This SAP will be finalized and approved before the clinical database lock. Any changes made to the SAP after the clinical database lock has occurred will be documented and discussed in the clinical study report for this study.

Sage Therapeutics, Inc. CONFIDENTIAL

## 3. STUDY OBJECTIVES

# 3.1. Primary Objective

The primary objective of this study is to assess the long-term safety and tolerability of SAGE-324.

# 3.2. Secondary Objective

The secondary objective of this study is to assess the long-term effect of SAGE-324 on other safety parameters.



Sage Therapeutics, Inc. CONFIDENTIAL

## 4. STUDY ENDPOINTS

# 4.1. Primary Endpoint

The primary endpoint of this study is the incidence of TEAEs.

# 4.2. Secondary Endpoints

The secondary endpoint(s) of this study are:

- The change from baseline in vital sign parameters
- The change from baseline in electrocardiogram (ECG) parameters
- The change from baseline in clinical laboratory parameters (eg, serum chemistry, hematology, coagulation, and urinalysis)
- Change from baseline in Epworth Sleepiness Scale (ESS) responses
- Physician Withdrawal Checklist (PWC-20) responses and total score
- Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) responses



Sage Therapeutics, Inc. CONFIDENTIAL

## 5. STUDY DESIGN

# 5.1. Overall Design

This study is an open-label study to evaluate the long-term safety and tolerability of SAGE-324 in participants with Essethtial Tremor (ET) who have completed the planned End of Treatment (EOT) Visit and who were not early terminated during the planned Treatment Period in another SAGE-324 study. This study includes a Screening Period of up to 28 days, a Treatment Period with weekly outpatient visits for the first 8 weeks, outpatient visits on Weeks 10, 12, 16, 20, and 24, and quarterly outpatient visits thereafter to the end of dosing, and a 14-day Follow-up Period. See the Schedule of Assessments (Appendix A) for the full list of study assessments and timings. The study is schematically presented in Figure 1.

Participants who have provided informed consent will undergo screening assessments up to

28 days prior to the planned day of dosing. Eligible participants will complete additional eligibility and baseline assessments.

Starting on Day 1, participants will self-administer on an outpatient basis a single dose of SAGE-324 once daily in the evening before bed, with a snack if bedtime is not within 2

hours of the evening meal. The dosing will start at 15 mg, and according to the dose escalation schedule provided in Figure 1 below, will be escalated to 60 mg starting on Day 43. If a participant experiences adverse events (AE) at any time during the Treatment Period that are considered by the investigator to be related to the investigational product (IP) and not tolerable, the investigator may reduce the dose of IP in 15 mg decrements, including during the initial dose escalation period. Administration of IP will be interrupted for 3 to 8 days before the initiation of the reduced dose.

During the Treatment Period, participants will return to the study center for safety, tolerability as specified in Appendix A. In addition, safety phone call study visits will be conducted as deemed appropriate by the investigator to review the current status of the participant. Participants will be trained in the use of software applications and devices necessary to complete questionnaires and/or self-rated study assessments.

The Treatment Period will continue for as long as the participant continues to self-administer SAGE-324 or until marketing authorization, projected to be up to approximately 5 years.

Follow-up visits will be conducted on an outpatient basis when participants have completed the Treatment Period. Participants will continue to complete questionnaires as indicated in Appendix A and will return to the clinic 3 (±3) days after the last dose of SAGE-324 for safety, tolerability at the End of Treatment (EOT) Visit.

Participants will return to the study center for an End of Study (EOS) Visit, 14 (±3) days after the last dose of SAGE-324.

Sage Therapeutics, Inc. CONFIDENTIAL





# 5.2. Sample Size and Power

The planned sample size is approximately 750 participants to be dosed and complete the study to contribute exposures to the safety database for SAGE-324 in accordance with ICH E1A guidelines.

## 5.3. Randomization

This is an open label study, hence no randomization is applicable.

# 5.4. Blinding and Unblinding

This is an open label study, hence no blinding is applicable.

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

# 6. MODIFICATIONS

# 6.1. Modifications from the Approved Clinical Study Protocol

There are no modifications in analysis specified in the clinical study protocol (version 4.0, dated 02 Nov 2023).

# 6.2. Modifications from the Approved Statistical Analysis Plan

This is the first version of the SAP for the final analysis.

# 6.3. Modifications from the Approved DMC Charter

Not Applicable.



# 7. ANALYSIS SETS

# 7.1. All Participants Set

The All Participants Set will include all participants who have given written informed consent.

# 7.2. Safety Set

The Safety Set is defined as all participants who administered at least one dose of SAGE-324.



Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

#### 8. STATISTICAL ANALYSIS

#### 8.1. General Considerations

All participant data, including those that are derived, that support the tables and figures will be presented in the participant data listings. Some data may be presented only in participant data listings, some may be presented with a corresponding table or figure; these will be indicated in relevant sections below.

For all safety analyses where applicable, baseline is defined as the last non-missing measurement prior to the first dose of IP. For scores that are made up of item scores, all item scores must come from the same visit to be considered as baseline for the overall score.

Continuous endpoints will be summarized with n, mean, standard deviation (SD), median, first and third quartiles (Q1, Q3), minimum (min), and maximum (max). The minimum and maximum will be reported with the same number of decimal places as the source (raw) data. Mean and median will be reported to 1 decimal place more than the source (raw) data and standard deviation will be reported to 2 decimal places more than the source (raw) data. Any values that require transformation to standard units (metric or SI) will be converted with the appropriate corresponding precision. In addition, change from baseline values will be calculated at each time point and summarized descriptively.

Categorical endpoints (eg, incidence of an adverse event) will be summarized using counts and percentages. Percentages will be presented to 1 decimal place unless otherwise specified.

Participants will be summarized according to treatment received. "By-visit" summaries are based on the last dose received before the specific evaluation. Adverse events summaries are based on the last dose received before the start of the AE. Note that it is possible for a participant to be counted under more than one dose in summaries. Since baseline is by definition before the first dose of IP, baseline values in listing will have no dose designation, and in summaries it will be presented under "Sage-324 Overall". For displays for which no such date applies, e.g. demographics, disease history, etc., the presentation will not be by dose group, but will be by aggregate SAGE-324 group.

# 8.2. Background Characteristics

## 8.2.1. Participant Disposition

The summary of disposition will use the All Participants Set and include number of participants who were screened, screen failed, successfully screened but did not dose, and successfully screened and dosed (overall and by previous study participation), and, using the number of participants who successfully screened and dosed as the denominator, the number and percentage of participants who completed treatment, who discontinued treatment (overall, by dose level, and by primary reason for discontinuing treatment), who completed the study, and who discontinued the study (overall and by primary reason).

Sage Therapeutics, Inc. CONFIDENTIAL

If a participant is rescreened because he/she has been a screen failure the first time, the status of the participant will be determined from the second screening. In the count of screened participants, such a participant will be counted only once.

A completer of the study is a participant with the study completion question answered 'Yes' on the End of Study / Study Disposition CRF page. A completer of treatment is a participant with the treatment completion question answered 'Yes' on the IP Completion / Discontinuation CRF page. The primary reason for discontinuing the study is provided in the respective CRF page.

The number of participants in each of the analysis sets will also be summarized and presented, using the All Participants Set. The reasons for participants being excluded from each analysis set will be listed (using All Participants) but not summarized.

#### 8.2.2. Protocol Deviations

Protocol deviations will be captured on eCRF and categorized by the study team as major and minor deviations. The major deviations will be summarized by type using the Safety Set. The minor deviations will be included in the listing but not summarized. The COVID-19 related protocol deviations will be summarized separately.

Inclusion/exclusion violations will be listed for All Participants (excluding screen failures) but not summarized.

# 8.2.3. Demographics and Baseline Characteristics

Demographic data (age, sex, race, and ethnicity), baseline characteristics (height, weight, BMI, dominant upper limb),

will be summarized with descriptive

statistics using the Safety Set.

Baseline subgroups will be summarized for the following categories:

- Race (Black or African American, White, Asian, Other)
- Sex (Female, Male)
- Age (<65, 65 to 80 years)</li>
- BMI (<18.5, 18.5 to <25, 25 to <30,  $\ge30$  kg/m<sup>2</sup>)

Listings will be provided for demographics, other baseline characteristics, and informed consent data.

Sage Therapeutics, Inc. CONFIDENTIAL

## 8.2.4. Medical/Surgical History

Medical/surgical history will be coded to Medical Dictionary for Regulatory Activities (MedDRA) terms, using Version 25, or higher. The MedDRA version will be included in the footnotes of related outputs. Medical/surgical history will be summarized using discrete summary statistics for each MedDRA System Organ Class (SOC) and Preferred Term (PT) using the Safety Set.

Age at ET diagnosis (years), age participant thinks ET started (years), years with ET diagnosis (age at baseline minus age at ET diagnosis), years since participant thinks ET started (age at baseline minus age when participant thinks ET started), tremor responsive to alcohol, past treatments for ET, and response to past treatment for ET will be summarized using the Safety Set. The data listing will also include reason for discontinuation from the past treatment.

The disease history will be summarized for the following categories:

- Age at ET diagnosis (<40 years, 40 to 60 years, >60 years)
- Age participant thinks ET started (<20 years, 20 to 40 years, >40 to 60 years, >60 years)
- Years with ET diagnosis (3 to <6 years, 6 to 10 years, >10 years)
- Years since participant thinks ET started (3 to <6 years, 6 to 10 years, >10 years)
- Tremor responsive to alcohol: Yes (Intermediate, Worked Well), No (No, a little), NA
- Past treatment for ET (Yes, No)
- Response to past treatment for ET: Yes (Intermediate, Worked Well), No (No, a little), Yes and No (denominator for percentages will be participants having past treatment for ET)

#### 8.2.5. Prior and Concomitant Medications

Medications will be recorded at each study visit and coded into drug class (anatomical therapeutic chemical [ATC] Level 2) and PT using World Health Organization-Drug dictionary (WHO-DD) Global B3 March 2022, or later.

All medications taken within 30 days prior to informed consent through the duration of the study (including start and end dates, route, dose/units, frequency, and indication) will be recorded on the electronic case report form (eCRF).

Those medications taken prior to the initiation of the IP will be denoted "Prior". Those medications taken prior to the initiation of the IP and continuing beyond the initiation of the IP or those medications started at the same time or after the initiation of the IP will be denoted "Concomitant". Note that medication taken before the initial dosing of IP and continued after the initial dosing will be categorized as a prior medication and separately as a concomitant medication.

Sage Therapeutics, Inc. CONFIDENTIAL

Medications will be flagged in the listing according to whether they are "Prior" or "Concomitant" as defined above. In the event of a missing start or stop date associated with a medication, only the classification (prior and/or concomitant) will be imputed using the algorithm described in <u>Appendix B</u>. Dates will not be imputed.

Prior and concomitant medications will be summarized separately using the Safety Set as the number and percentage of participants with each medication at both the ATC and PT levels. Concomitant procedures will be listed with SOC/PT, but not summarized.

# 8.2.6. Investigational Product Exposure

Total investigational product exposure (in mg) is defined as the total mg of SAGE-324 that was taken during the study. If a participant skips a dose on any of the days, the dose taken is 0 mg.

Total exposure duration to SAGE-324 (in days) is defined as (date of last dose – date of first dose + 1). Note that this does not exclude days when the dose has been missed.

Planned exposure for participants with no unscheduled dose reductions/increases is defined as the sum of:

- 14 days of treatment (Day 1 through Day 14) times 15 mg
- 14 days of treatment (Day 15 through Day 28) times 30 mg
- 14 days of treatment (Day 29 through Day 42) times 45 mg
- Number of days from Day 43 to end of treatment, inclusive, times 60 mg

If a participant has an unscheduled dose reduction/increase, or dose reductions/increases, planned exposure will be as indicated until the point of the first unscheduled reduction/increase. Planned exposure from the point of the first unscheduled reduction/increase will be the assigned dose times the number of days from the date of the reduction/increase (inclusive) to the date of the next reduction/increase (exclusive) or the date of end of treatment (inclusive). Planned exposure for any additional unscheduled reductions/increases will be handled in a similar manner as the assigned dose times the number of days from the date of the reduction/increase (inclusive) to the date of the next reduction/increase (exclusive) or the date of end of treatment (inclusive).

Percent of the planned exposure received is defined as the total investigational product exposure, divided by planned exposure, times 100.

Total investigational product exposure, total exposure duration, and percent of planned exposure received will be summarized using the Safety Set. The number and percentage of participants with percent of planned exposure received <80%, 80% to <100%, and ≥100% will be summarized. Total exposure duration (over all doses taken) will also be summarized by dose at time of treatment discontinuation using the Safety Set.

Sage Therapeutics, Inc. CONFIDENTIAL

## 8.2.7. Investigational Product Adherence

IP adherence (%) is defined as the number of tablets taken, divided by the number of tablets planned to be taken, times 100. Number of tablets planned to be taken will be derived using an algorithm identical to that used for the derivation of planned exposure, but with the assigned dose replaced with the number of assigned tablets (15 mg = 1 tablet per day, 30 mg = 2 tablets per day, 45 mg = 3 tablets per day, 60 mg = 4 tablets per day).

Total tablets taken and IP adherence will be summarized descriptively using the Safety Set. Number and percentage of participants with IP adherence in categories <75%, 75 to 100%, >100% will be provided.



Sage Therapeutics, Inc. CONFIDENTIAL



Sage Therapeutics, Inc. CONFIDENTIAL



Statistical Analysis Plan Methods Version 1.0 22Oct2024

Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

Sage Therapeutics, Inc.

Sage Therapeutics, Inc. CONFIDENTIAL



Sage Therapeutics, Inc. CONFIDENTIAL

# 8.4. Safety Analysis

Safety and tolerability of SAGE-324 will be assessed based on TEAEs, changes from baseline in clinical laboratory evaluations, 12-lead ECGs, and vital signs, C-SSRS, PWC-20, and ESS. Safety data will be listed by participant.

For safety summary tables, the safety endpoints evaluated at scheduled visits are taken as done and nominal visit will be summarized as scheduled visits. For multiple values from the specific visit window, the choice of the visit record will be following the same rule as described in <u>Section 8.3.2</u>.

All safety summaries will be prepared by dose level and overall for the Safety Set. See <u>Table</u> 4 for details on how safety endpoints will be presented.

**Table 4: Presentation of Safety Endpoints** 

| Safety<br>Evaluation | Incidence | Raw Value | Change from<br>Baseline | Abnormality | Derived PCS values |
|---|---|---|---|---|---|
| TEAEs | X | * | | | |
| Vital Signs | | X, * | X | | X, * |
| 12-lead ECG | | X, * | X | X, * | X, * (QTcF<br>only) |
| Safety Labs<br>(Chemistry,<br>Hematology,<br>Urinalysis) | | X, * | X | X, * | X, * |
| ESS | X | * | X | | |
| PWC-20 | X | * | | | |
| C-SSRS | X | * | X | | |

X = Safety Assessment will be summarized in tables

Note: PCS = Potentially Clinically Significant.

# 8.4.1. Adverse Events

Adverse events will be coded using MedDRA Version 25 or higher. In the event of a missing/incomplete start or stop date associated with an adverse event, only the treatment-emergence will be imputed using the algorithm described in <a href="Appendix B">Appendix B</a>. Dates will not be imputed.

A TEAE is defined as an AE with onset at or after the first dose of IP (SAGE-324). Summary tables of AEs will include TEAEs only and will summarize data using the Safety Set participants overall and by dose level taken immediately prior to the AE onset.

An overall adverse event summary table will be presented for TEAEs and will include the number and percent of participants experiencing at least one:

- TEAE
- Maximum severity of TEAE (mild TEAE, moderate TEAE, severe TEAE)

<sup>\* =</sup> Safety Assessment will be presented in individual participant data listings

Sage Therapeutics, Inc. CONFIDENTIAL

- TEAE leading to dose interruption
- TEAE leading to dose reduction
- TEAE related to IP
- TEAE leading to IP discontinuation
- TEAE leading to study discontinuation
- Serious TEAE
- Serious TEAE related to IP
- Serious TEAE leading to IP discontinuation
- Serious TEAE leading to study discontinuation
- TEAE resulting in death

The incidence of TEAEs will be summarized by System Organ Class (SOC) and Preferred Term (PT). In addition, summaries will be provided by maximum severity (mild < moderate < severe) and by maximum relationship (related > not related) to IP. Any TEAEs leading to IP discontinuation, any TEAE leading to study discontinuation, and any treatment-emergent SAEs will also be summarized, sorted by descending frequency in SOC and PT.

Participants will be counted only once within each SOC and PT at the maximum severity in the following order: severe, moderate, and mild. Participants will be counted only once within each SOC and PT at the strongest relationship to IP in the following order: related, not related to IP. An AE with missing severity will be considered as 'severe', and with missing relationship to IP will be considered as 'related' for the purposes of summarizing these data.

The incidence of TEAEs and treatment-emergent SAEs will also be presented in order of decreasing frequency by PT.

All AEs (including those with onset before the start of IP) through the end of the study will be listed. In addition, separate listings containing individual participant AE data for all deaths, SAEs, AEs leading to IP discontinuation, and AEs leading to study discontinuation will be provided.

## 8.4.2. Clinical Laboratory

All statistical analyses of laboratory values will be performed using SI units. The following parameters are mentioned in the protocol, hence will be summarized; any other parameters for which data are reported will be listed but not summarized.

## Biochemistry:

- Renal Panel: glucose, calcium, phosphorus, blood urea nitrogen, creatinine, sodium, potassium, chloride, total carbon dioxide content
- Hepatic Panel: albumin, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, direct bilirubin, indirect bilirubin, alkaline phosphatase, total protein, lactate dehydrogenase, gamma glutamyl transferase, creatine kinase (MB and MM)

Sage Therapeutics, Inc. CONFIDENTIAL

 Other: total lipid profile, creatine phosphokinase, thyroid stimulating hormone (TSH), alcohol level, HbA1c

## Coagulation:

 Activated partial thromboplastin time, prothrombin time, and international normalized ratio

#### Hematology:

 Red blood cell (RBC) count, hemoglobin, hematocrit, white blood cell count with differential, platelet count, and if RBC indices are abnormal, reflex RBC morphology is indicated

#### Urinalysis:

 Protein, glucose, pH, blood, leukocytes, leukocyte esterase, urobilinogen, bilirubin, ketones, nitrite, myoglobin

Some numeric lab values may be reported as '<n.n' or '>n.n'; these will be analyzed in the summary statistics as n.n/2 and n.n, respectively. For example, triglycerides recorded as "<0.50" mmol/L would be analyzed as 0.25 mmol/L and potassium recorded as ">6.0 mmol/L" would be analyzed as 6.0 mmol/L.

All by-visit laboratory summary tables will present results for the Safety Set participants overall, and by dose level received prior to the given evaluation. For summarization of incidence data any time post-baseline, participant data will be summarized according to the last dose received when a particular criterion was met (thus, a participant may contribute data under more than one dose if a criterion was met post-baseline while taking different doses).

Continuous hematology, chemistry, coagulation, and urinalysis results (raw and change from baseline) will be summarized at each scheduled time point. Categorical urinalysis results will be summarized by frequencies and percentages at each scheduled time point. The number and percentage of participants with shift from baseline based on the laboratory normal ranges provided by the laboratory will be tabulated at each scheduled visit.

Any laboratory value considered clinically significant by the investigator is captured as an adverse event.

The number and percentage of participants with potentially clinically significant (PCS) values at any time after IP administration (including unscheduled visits) will be summarized for the hematology, chemistry, and coagulation parameters defined in <u>Table 5</u>, <u>Table 6</u>, and <u>Table 7</u>, respectively. PCS values for each scheduled visit and end-of-treatment and end-of-study values will also be provided. These summaries will be done using the Safety Set, overall for SAGE-324 as well as by dose level.

Liver function tests will be monitored closely; PCS values (<u>Table 8</u>) will be summarized using the Safety Set for incidence any time post-baseline for these PCS thresholds (for conditions involving more than one parameter, the results need to be from the same timepoint).

Sage Therapeutics, Inc. CONFIDENTIAL

Chemistry, hematology, coagulation, and urinalysis data will be listed with the values outside the normal ranges and PCS criterion flagged. Blood cell morphology and microscopy test results will be listed when available but not summarized. Virus serology, pregnancy tests, and urine drugs of abuse data will be listed but not summarized.

Table 5: Potentially Clinically Significant Values for Hematology

| Laboratory Parameter | Sex | Units | Criteria for PCS Values (Observed values) | |
|---|---|---|---|---|
| | | | High | Low |
| Hemoglobin | Male | g/L | >185 | <115 |
| | Female | g/L | >170 | <100 |
| Hematocrit | Male | Fraction of 1 | >0.55 | < 0.385 |
| | Female | Fraction of 1 | >0.49 | < 0.345 |
| Platelet count | | 10^9/L | >600 | <125 |
| White blood cell | | 10^9/L | >15 | <2.5 |
| Basophils | | 10^9/L | >0.5 | NA |
| Eosinophils | | 10^9/L | >1.5 | NA |
| Neutrophils | | 10^9/L | NA | <1.5 |
| Lymphocytes | | 10^9/L | >6.0 | <0.5 |
| Monocytes | | 10^9/L | >1.4 | NA |

Table 6: Potentially Clinically Significant Values for Chemistry

| Laboratory Parameter | Units | Criteria for PCS Values (Observed values) | |
|---|---|---|---|
| _ | | High | Low |
| Albumin | g/L | >70 | <28 |
| Blood urea nitrogen | mmol/L | >10.71 | NA |
| Calcium | mmol/L | >2.75 | <2.0 |
| Chloride | mmol/L | >120 | <90 |
| Creatinine | mmol/L | >3xULN or >3x Baseline | |
| Gamma Glutamyl Transferase | | >3xULN | |
| Glucose | mmol/L | >13.9 | <2.8 |
| Sodium | mmol/L | >150 | <132 |
| Potassium | mmol/L | >5.4 | <3.3 |
| Protein | g/L | | <45 |
| Bicarbonate | mmol/L | >34 | <18 |
| Chloride | mmol/L | >120 | <90 |
| Phosphorus | mmol/L | >1.94 | < 0.61 |
| Liver Function Tests (LFT) | | | |
| Bilirubin | μmol/L | >2xULN | |
| Aspartate Aminotransferase | U/L | >3xULN | |
| Alanine Aminotransferase | U/L | >3xULN | |
| Alkaline Phosphatase | U/L | >1.5xULN | |

Table 7: Potentially Clinically Significant Values for Coagulation

| Parameter | Potentially Clinically Significant Values |
|---|---|
| Prothrombin time (PT) | >=1.11 x ULN |
| Activated partial thromboplastin time (aPTT) | >1.5 x ULN |

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

Table 8: Potentially Clinically Significant Values for Liver Function Tests

| Parameter | Potentially Clinically Significant Values |
|---|---|
| Alanine Aminotransferase | >3xULN, >5xULN, >10xULN |
| Aspartate Aminotransferase | >3xULN, >5xULN, >10xULN |
| Alanine Aminotransferase OR | >3xULN, >5xULN, >10xULN |
| Aspartate Aminotransferase | |
| Alkaline Phosphatase | >1.5xULN, >2xULN |
| Total Bilirubin >1.5xULN, >2xULN | |
| Total Bilirubin > 2xULN AND (Alanine Aminotransferase OR Aspartate Aminotransferase | |
| >3xULN), any time postbaseline, do not need to be at the same visit | |
| Potential Hy's Law: [Total Bilirubin >=2xULN AND Alkaline Phosphatase <2xULN, measured at | |
| the same visit] AND [(Alanine Aminotransferase OR Aspartate Aminotransferase >3xULN) AND | |
| Alkaline Phosphatase <2xULN, measured at the same visit], two conditions at any time | |
| postbaseline, do not need to be at the same visit | |

## 8.4.3. Electrocardiogram

All by-visit ECG summary tables will present results for Safety Set participants overall, and also by dose level received prior to the evaluation. For summarization of incidence any time post-baseline, participant data will be summarized according to the last dose received when a particular criterion was met (thus, a participant may contribute data under more than one dose if a criterion was met post-baseline while taking different doses). Last value on treatment and last value on study will be summarized under the dose level last received.

The average of any multiple values collected at one visit will be used for summarization of continuous variables, including baseline ECG values. For each ECG measurement (heart rate and PR, QRS, QT, and QTcF intervals), the observed value at each scheduled visit and change from baseline at each scheduled visit will be provided. This summary will also include last values on treatment and on study. Last value on treatment is defined as the last post-baseline value between first dose of IP (exclusive) and up to last dose of IP + 1 day (inclusive). Last value on study is defined as the last post-baseline value after the first dose of IP.

In addition, the number and percentage of participants with PCS and potentially clinically significant change (PCSC) values will be summarized by scheduled timepoint and for any time post-baseline, including last value on treatment and last value on study. Individual values of QTcF will be used for PCS determination rather than the average of multiple values collected at one visit. Potentially clinically significant values will be identified for ECG parameters as outlined in <u>Table 9</u>.

A shift table of overall ECG interpretation from baseline to scheduled post-baseline visits will be presented for the following categories: 'Normal', 'Abnormal, Not Clinically Significant', and 'Abnormal, Clinically Significant'. The shift table will be presented by visit – overall and by dose level.

Clinically significant abnormal findings will be reported as adverse events. The average of any multiple values collected at one visit of each parameter will be included in the data listing.

Sage Therapeutics, Inc. CONFIDENTIAL

Table 9: Potentially Clinically Significant Values for QTcF

| Units | Criteria for PCS Values<br>(Observed Values) | | Criteria for PCSC Values<br>(Change from Baseline) | |
|---|---|---|---|---|
| | High Low | | Increase | Decrease |
| msec | >450 msec and ≤480msec<br>>480 msec and ≤500msec<br>>500 msec | NA | >30 msec and ≤60 msec<br>>60 msec | NA |

# 8.4.4. Vital Signs

All by-visit vital sign summary tables will present results for Safety Set participants overall, and also by dose level received prior to the evaluation. For summarization of incidence at any time post-baseline, participant data will be summarized according to the last dose received when a particular criterion was met (thus, a participant may contribute data under more than one dose if a criterion was met post-baseline while taking different doses).

Vital sign results (systolic and diastolic blood pressure [mmHg], pulse pressure (mmHg), body temperature [°C], heart rate [beats per minute or bpm], and respiratory rate [breaths per minute]) and changes from baseline will be summarized by scheduled visit – overall and by dose level. Pulse pressure is defined as [systolic blood pressure - diastolic blood pressure].

Potentially clinically significant values will be identified for vital sign parameters as outlined in <u>Table 10</u>. For any post-baseline visit, potentially clinically significant values will be summarized by visit.

Any vital sign results considered clinically significant by the investigator will be captured as adverse events.

Sage Therapeutics, Inc. CONFIDENTIAL

Table 10: Potentially Clinically Significant Values for Vital Sign Parameters

| Vital Sign | Units | Criteria for PCS Values<br>(Observed values) | | Criteria for PCSC<br>values (Change from<br>Baseline values) | |
|---|---|---|---|---|---|
| | | High | Low | Increase | Decrease |
| Heart rate<br>(supine and standing) | Beats/min | >120 | <40 | | |
| Systolic Blood Pressure<br>(supine and standing) | mmHg | >180 | <90 | ≥30 | ≥30 |
| Diastolic Blood pressure<br>(supine and standing) | mmHg | >110 | <50 | ≥20 | ≥20 |
| Supine - Standing<br>Systolic Blood Pressure | mmHg | ≥20 | | | |
| Supine – Standing<br>Diastolic Blood Pressure | mmHg | ≥10 | | | |
| Orthostatic hypotension:<br>supine – standing SBP and | mmHg | SBP ≥20 and<br>DBP ≥10 | | | |
| DBP | | SBP ≥20 or DBP<br>≥10 | | | |

# 8.4.5. Physical Examination

The occurrence of a physical examination and the date and time, along with the results of the mental status exam and the abbreviated neurological exam are collected. These will be presented in individual participant data listings only using the Safety Set. After screening, any clinically significant abnormal findings in physical examinations will be reported as AEs.

#### 8.4.6. Columbia Suicide Severity Rating Scale (C-SSRS)

All by-visit C-SSRS summary tables will present results for Safety Set participants overall, and also by dose level received prior to the given visit. For summarization of incidence data any time post-baseline, Safety Set participant data will be summarized according to the dose received immediately prior to the evaluation (thus, a participant may contribute data under more than one dose if a criterion was met post-baseline while taking different doses).

Suicidality data collected on the C-SSRS is collected during the clinic visits at Screening and post-baseline visits. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation with numeric rating for the severity (from 1 to 5 with 5 being the most severe) and behavior (from 6 to 10 with 10 being most severe). The "Baseline/Screening" C-SSRS form will be completed at screening (lifetime history and past 24 months). The "Since Last Visit" C-SSRS form will be completed at all subsequent visits.

The categorical outcomes of C-SSRS with binary response ("Yes"/ "No") include: Suicidal ideation with 5 being the worst:

1: wish to be dead

Sage Therapeutics, Inc. CONFIDENTIAL

- 2: non-specific active suicidal thoughts
- 3: active suicidal ideation with any methods (not plan) without intent to act
- 4: active suicidal ideation with some intent to act, without specific plan
- 5: active suicidal ideation with specific plan and intent

Suicidal behavior with 10 being the worst:

- 6: preparatory acts or behavior
- 7: aborted attempt
- 8: interrupted attempt
- 9: actual attempt
- 10: completed suicide

Suicidal behavior is considered worse than suicidal ideation. The participant's non-suicidal self-injurious behavior is also assessed separately as part of C-SSRS:

11: self-injurious behavior without suicidal intent

Baseline for each question is defined as the worst of the assessments done before the first dose of IP, excluding the lifetime version. This will typically include the 'past 24-month' version from screening and 'since last visit' version from Day 1, as well as any unscheduled visits done before the first dose of IP; any 'Yes' response will make the baseline value as 'Yes'.

The number and percentage of participants with at least one response of 'Yes' to any C-SSRS suicidal ideation or suicidal behavior item, as well as for participant's non-suicidal self-injurious behavior, will be summarized by visit.

Change from baseline for C-SSRS will be assessed using shift tables. Summary of shift from baseline in C-SSRS suicidal ideation and suicidal behavior will be presented for the categories "no suicidal ideation/behavior", "suicidal ideation", and "suicidal behavior" for each scheduled assessment time point. If the answer to all 5 assessments in suicidal ideation and all 5 assessments in suicidal behavior is 'No', then the category for the table is considered as 'No suicidal ideation/behavior'. If any of the assessments in suicidal behavior are 'Yes', the category is considered as 'Suicidal behavior are 'Yes' but all assessments in suicidal behavior are 'No', the category is considered as 'Suicidal ideation'.

In addition, a summary of shift in suicidal ideation from baseline maximum rank score for any time post-baseline maximum rank score will be presented. Maximum score 0 refers to all 'No' for all assessments in the desired period for all 5 questions on suicidal ideation.

## 8.4.7. Physician Withdrawal Checklist (PWC-20)

The PWC-20 is a shorter version of the Penn Physician Withdrawal Checklist based on the 20 items that provided the best differentiation from placebo in previous trials. The PWC-20

Sage Therapeutics, Inc. CONFIDENTIAL

is made up of a list of 20 symptoms (eg, loss of appetite, nausea-vomiting, diarrhea, anxiety-nervousness, irritability) that are rated on a scale of 0 (not present) to 3 (severe) (<u>Rickels 2008</u>). The PWC-20 will be used to monitor for the presence of potential withdrawal syndrome following discontinuation of SAGE-324.

Summarization of PWC-20 data will be presented using the Safety Set — overall and by dose last received immediately prior to the evaluation. Descriptive statistics for the total PWC-20 score will be presented at End of Treatment (defined as the first available assessment after the last dose of study within 1 day of last dose) and End of Study. The change from End of Treatment to End of Study in PWC-20 total score will be provided. The number and percentage of participants with each PWC-20 item and reporting severe on a PWC-20 item will be presented at each visit. Descriptive statistics for the number of PWC-20 items and the number of severe PWC-20 items experienced at each visit will also be presented.

#### 8.4.8. Epworth Sleepiness Scale (ESS)

The ESS is a quick, 8-item, self-administered questionnaire where participants rate, on a 4-point scale of 0 (no chance of dozing) to 3 (high chance of dozing), their usual chances of dozing off or falling asleep while engaged in 8 different activities. The total ESS score estimates the participant's average sleep propensity, across a range of activities in their daily lives (Johns 2002).

All by-visit ESS summary tables will present results using the Safety Set – overall, and also by dose last received immediately prior to the evaluation. Descriptive statistics for each of the 8 individual items (continuous and by categorical response) at each scheduled visit, the total ESS score at each scheduled visit, and change from baseline in the total ESS score at each postbaseline visits will be presented. The number and percentage of participants with a total ESS score of 0, no chance of dozing off, will also be presented at each visit.

#### 8.4.9. Other Safety Analysis

Not applicable.



Not applicable.

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Sage Therapeutics, Inc. Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) CONFIDENTIAL

# 9. SUMMARY OF INTERIM AND DMC ANALYSES

# 9.1. Interim Analysis

Not applicable.

# 9.2. DMC Analysis

Not applicable.

Sage Therapeutics, Inc. CONFIDENTIAL

## 10. REFERENCES

Deuschl G, Raethjen J, Hellriegel H, et al. Treatment of patients with essential tremor. Lancet Neurol. 2011;10(2):148-61.



Hopfner F, Haubenberger D, Galpern WR, et al. Knowledge gaps and research recommendations for essential tremor. Parkinsonism Relat Disord. 2016;33:27-35.

Johns MW. Sleep propensity varies with behaviour and the situation in which it is measured: the concept of somnificity. J Sleep Res. 2002;11:61-7.

Koller WC, Busenbark K, Miner K. The relationship of essential tremor to other movement disorders: report on 678 patients. Essential Tremor Study Group. Ann Neurol. 1994;35(6):717-23.

Koller WC, Vetere-Overfield B. Acute and chronic effects of propranolol and primidone in essential tremor. Neurology. 1989;39(12):1587-8.

Louis ED, Ottman R. How many people in the USA have essential tremor? Deriving a population estimate based on epidemiological data. Tremor Other Hyperkinet Mov (N Y). 2014;4:259.

NIH. Genetics Home Reference: Essential Tremor. Bethesda, MD: U.S. Department of Health and Human Services, National Institutes of Health. Published 15 Oct 2019. Available from: https://ghr.nlm.nih.gov/condition/essential-tremor.

Olanow CW. Hyperkinetic Movement Disorders: Essential Tremor. Harrison's Principles of Internal Medicine. 17 ed. New York, NY: McGraw Hill; 2008. p. 2560.

Posner K, Brown GK, Stanley B, et al. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011;168(12):1266-77.

Rajput AH, Rajput A. Medical treatment of essential tremor. J Cent Nerv Syst Dis. 2014;6:29-39.

Rickels K, Garcia-Espana F, Mandos LA, Case GW. Physician Withdrawal Checklist (PWC-20). J Clin Psychopharmacol. 2008;28(4):447-451.

Wyeth. Inderal (propranolol hydrochloride) [package insert]. Philadelphia, PA; 2010.

Sage Therapeutics, Inc. CONFIDENTIAL

Zappia M, Albanese A, Bruno E, et al. Treatment of essential tremor: a systematic review of evidence and recommendations from the Italian Movement Disorders Association. J Neurol. 2013;260(3):714-40.
Sage Therapeutics, Inc. CONFIDENTIAL

# 11. LIST OF APPENDICES

Docusign Envelope ID: 1171D0B2-DF24-43FC-AB7E-BD0FEEFD3DF8

# APPENDIX A. SCHEDULE OF ASSESSMENTS

Docusign Envelope ID: 1171D0B2-DF24-43FC-AB7E-BD0FEEFD3DF8

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023)

| Assessment | Screening | | | | I | Treatment Period | Po | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -28 to -1 | 1 | 90 | 15 | 22 | 29 | 36 | 43 | 90 | 57 |
| Window (Days) | | | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 |
| Informed consent | X | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | |
| Demographics | X | | | | | | | | | |
| Medical history | X | | | | | | | | | |
| Pregnancy test | X<br>(serum; all<br>women) | X<br>(urine; WOCBP<br>only) | | | | X<br>(urine;<br>WOCBP only) | | | | X<br>(urine;<br>WOCBP only) |
| FSH (postmenopausal<br>women only) | x | | | | | | | | | |
| Drug screen | X | × | | | | | | | | |
| Complete physical examination, including metrological examination including MSE* | х | | | | | | | | | |
| Body height | x | | | | | | | | | |
| Body weight | X | | | | | | | | | |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X |
| 12-Lead ECG <sup>c</sup> | X | x | | | | | | x | | |
| Chemistry/hematology/<br>coagulation/urinalysis <sup>d</sup> | X | x | x | x | | x | | x | | × |

Sage Therapeutics, Inc. CONFIDENTIAL

Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) Statistical Analysis Plan Methods Version 1.0 22Oct2024

| Assessment | Screening | | | | Ţ | Treatment Period | poi | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -28 to -1 | I | 8 | 15 | 22 | 29 | 36 | 43 | 50 | 57 |
| Window (Days) | | | ±2 | ±2 | ∓2 | ∓2 | ±2 | ±2 | ±2 | ±2 |
| C-SSRS<br>("Screening/Baseline"<br>form) | X | | | | | | | | | |
| C-SSRS<br>("Since Last Visit" form) | | x | x | x | x | x | x | x | x | × |
| ESS | X | X | × | X | x | X | X | X | X | × |
| Participant trainings | x | x | | | | | | | | |
| Dispense SAGE-324h | | X | × | × | × | x | x | × | × | × |
| SAGE-324 accountability | | | X | X | X | X | X | X | X | × |
| SAGE-324 administration | | | | | Administer | Administered once daily before bed | before bed | | | |
| AEs/SAEs | | 134 | | | | X | | | | |
| Prior medication and<br>history <sup>d</sup> | x | | | | | | | | | |
| Concomitant medication | x | | | | | X | | | | |
| Alcohol, nicotine products, and dietk | | | | | | × | | | | |

Abbreviations: AE = adverse event; C-SSRS = Columbia-Suicide Severity Rating Scale; ECG = electrocardiogram; ESS = Epworth Sleepiness Scale; ET essential tremor; FSH = follicle stimulating hormone; ICF = informed consent form; IP = investigational product; MSE = mental state examination; SAE = serious adverse event;

clinical laboratory WOCBP = women of childbearing potential.

during clinic visits is vital signs, ECG, blood sample collection for Note: The suggested order of assessments during clinic visits is vital signs, assessments, and questionnaires.

38

Sage Therapeutics, Inc. CONFIDENTIAL

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) <sup>a</sup> Complete physical examination and a comprehensive neurological examination, including MSEs, should be performed at Screening and as clinically necessary (see Section 12.1.3). Targeted physical and neurological examinations should be performed at other times as indicated by AEs.

standing blood pressure and heart rate will be collected in triplicate at least 15 minutes apart., measured after the participant has been in the supine position participant has been in the supine position for at least 5 minutes and then repeated approximately 1 and 3 minutes after standing. On Day 1, supine and b Vital signs comprise heart rate, respiratory rate, temperature, and blood pressure. Systolic and diastolic blood pressure are to be measured after the participant has been supine for at least 5 minutes prior to the measurement. Orthostatic blood pressure and heart rate will also be measured after the for at least 5 minutes and then repeated 1 minute and 3 minutes after standing. Respiratory rate and temperature are collected once on Day 1.

<sup>e</sup> ECGs will be collected and read locally. All ECGs must be performed after the participant has been in a supine position for at least 5 minutes.

(biochemistry) at Screening and at additional timepoints at the discretion of the investigator. A serum sample for blood alcohol level will be collected at d Chemistry, hematology, coagulation, and urinalysis at Screening and at all additional timepoints. Myoglobin (urinalysis) and serum creatine kinase Screening and all additional timepoints. HbA1c will be collected at Screening.

At the discretion of the investigator, clinical laboratory assessments from another SAGE-324 study may be used to determine eligibility for this study if within 28 days of Day 1.

8 Participants will be trained by study personnel on the use of software applications, IP diary, and devices necessary for the conduct of the study

and not tolerable, the investigator may reduce the dose of IP in 15 mg decrements, including during the initial dose escalation period. Self-administration of daily starting on Day 43. If a participant experiences AEs that are considered at any time in the Treatment Period by the investigator to be related to the IP h Participants will self-administer orally 15 mg SAGE-324 on Day 1 to Day 14, 30 mg on Day 15 to Day 28, 45 mg on Day 29 to Day 42, and then 60 mg IP will be interrupted for 3 to 8 days before the initiation of the reduced dose.

Participants will self-administer orally on an outpatient basis a single dose of SAGE-324 once daily in the evening before bed, with a snack if bedtime is not within 2 hours of the evening meal.

Including all medications and supplements taken within the 30 days prior to signing the ICF through the first dose of SAGE-324, as well as a complete history of all treatments for ET since the year of diagnosis.

<sup>k</sup> Alcohol, nicotine use and diet will be collected to ensure compliance with IC#9, IC#10, and EC#14, respectively.

Docusign Envelope ID: 1171D0B2-DF24-43FC-AB7E-BD0FEEFD3DF8

Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) Statistical Analysis Plan Methods Version 1.0 22Oct2024

Treatment Period Week 10 to Week 24

| Study Week 10 12 16 20 24 Window (Weeks) ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 ±1 </th <th> 12</th> <th>Assessment</th> <th></th> <th></th> <th>Treatment Period</th> <th></th> <th></th> | 12 | Assessment | | | Treatment Period | | |
|---|---|---|---|---|---|---|---|
| Manacy test | ±1 | Study Week | 10 | 12 | 16 | 20 | 24 |
| Notice N | X X X X X X X X X X X X X | Window (Weeks) | 11 | 11 | 11 | 17 | 11 |
| Signs Sacoultability Sacoultabilit | X X X X X X X X X X X X X X X X X X X | Pregnancy test | X (urine; WOCBP only) | | X<br>(urine; WOCBP only) | | X<br>(urine; WOCBP only) |
| signs b ead ECG* X X X X mistry/hematology/ coagulation/urnalysis4 X X X X RS X X X X X ce Last Visit* form) X X X X X ce Last Visit* form) X X X X X cuse SAGE-324* X X X X X X E-324 accountability X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X < | X X X X X X X X X X X X X X X X X X X | Complete physical examination, including neurological examination including MSE <sup>a</sup> | | x | | | x |
| sed ECG* X X X nistry/hematology/ coagulation/urinalysis <sup>d</sup> X X X X sRS X X X X X src Last Visit" form) X X X X X X ense SAGE-324* X X X X X X X X E-324 accountability X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | Vital signs <sup>b</sup> | x | x | x | x | x |
| instry/hematology/ coagulation/urmalysis <sup>d</sup> X X X X ice Last Visit" form) X X X X ice Last Visit" form) X X X X cuse SAGE-324f X X X X ice Last Visit" form) X X X X ice 2324 administration* X X X X | X X X X X X X X X X X X X X X X X X X | 12-Lead ECG <sup>c</sup> | | x | | | x |
| RS X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | Chemistry/hematology/ coagulation/urmalysis <sup>d</sup> | | x | | | x |
| case SAGE-324f X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | C-SSRS<br>("Since Last Visit" form) | × | × | × | × | × |
| E-324 accountability X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | X X X X X X X Administered once dail Administered once dail X X X X X X X X ECG blood cample coll | | | | | | |
| X X X X nf X X X Administered once daily before bed X X X X X X X | X X X Administered once daily X X X X X X X X Rating Scale: ECG blood cample coll | ESS | X | X | X | X | X |
| Administered once daily before bed X Administered N X X X | Administered once daily Administered once daily X X X Sale: ECG = electrocardic | Dispense SAGE-324f | x | X | x | x | X |
| D <sub>2</sub> | Administered once dail X X Rating Scale: ECG = electrocardic | SAGE-324 accountability | x | x | x | x | X |
| | X Rating Scale: ECG = electrocardic | SAGE-324 administration <sup>‡</sup> | | Admi | nistered once daily bel | fore bed | |
| | X Rating Scale: ECG = electrocardic | AEs/SAEs | | | x | | |
| | Rating Scale: ECG = electrocardic | Concomitant medication | | | X | | |
| | ECU, plood sample collection for | Note: The suggested order of assessments during clinic visits is vital signs, | clinic visits is vital sig | | blood sample collecti | on for | Il laboratory |

assessments, and questionnaires.

Docusign Envelope ID: 1171D0B2-DF24-43FC-AB7E-BD0FEEFD3DF8

Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023) Statistical Analysis Plan Methods Version 1.0 22Oct2024

Sage Therapeutics, Inc. CONFIDENTIAL

<sup>a</sup> Complete physical examination and a comprehensive neurological examination, including MSEs, should be performed as clinically necessary (see Section

b Vital signs comprise heart rate, respiratory rate, temperature, and blood pressure. Systolic and diastolic blood pressure are to be measured after the participant has been supine for at least 5 minutes prior to the measurement. Orthostatic blood pressure and heart rate will also be measured after the participant has been in the supine position for at least 5 minutes and then repeated approximately 1 and 3 minutes after standing. (2.1.3). Targeted physical and neurological examinations should be performed as indicated by AEs.

(biochemistry) at Screening and at additional timepoints at the discretion of the investigator. A serum sample for blood alcohol level will be collected at d Chemistry, hematology, coagulation, and urinalysis at Screening and at all additional timepoints. Myoglobin (urinalysis) and serum creatine kinase ECGs will be collected and read locally. All ECGs must be performed after the participant has been in a supine position for at least 5 minutes. Screening and all additional timenoints. HgA1c will be collected at Week 12 and Week 24. If a participant experiences AEs at any time during the Treatment Period that are considered by the investigator to be related to the IP and not tolerable, the investigator may reduce the dose of IP in 15 mg decrements. Self-administration of IP will be interrupted for 3 to 8 days before the initiation of the reduced

<sup>8</sup> Participants will self-administer on an outpatient basis a single dose of SAGE-324 once daily in the evening before bed, with a snack if bedtime is not within 2 hours of the evening meal.

Docusign Envelope ID: 1171D0B2-DF24-43FC-AB7E-BD0FEEFD3DF8

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023)

Month 9 to Follow-up Period

| Mouth 9 Month 12 Month 15 Month 18 Month 24 to EOT | Assessment | | | Treatme | Treatment Period | | | Follow- | Follow-up Period |
|---|---|---|---|---|---|---|---|---|---|
| dow (Weeks) ±2 | Study Month | Month 9 | Month 12 | Month 15 | Month 18 | Month 21 | Month 24 to<br>Month 60<br>(Every<br>3 Months) | EOT 3 (±3) days after last dose of SAGE-324 | EOS 14 (±3) days after last dose of SAGE-324 |
| MoCBP only) WOCBP only) | Window (Weeks) | #5 | # | 77 | #5 | 77 | 77 | | |
| Plete physical | Pregnancy test | X<br>(urine;<br>WOCBP only) | | | | | X<br>(urine; WOCBP<br>only) | | X<br>(urine; WOCBP<br>only) |
| rweight b X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Complete physical examination including MSE <sup>a</sup> | × | × | × | × | × | x | × | × |
| signs <sup>c</sup> X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Body weight b | | × | | | | X | | х |
| ead ECG <sup>4</sup> X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Vital signs c | X | X | X | X | X | X | X | X |
| Nistry/hematology/ | 12-Lead ECG <sup>d</sup> | X | X | X | X | x | X | X | х |
| RS X X X X X X x = 20 x x x x x x x x = | Chemistry/hematology/<br>coagulation/urnalysis* | × | × | × | x | × | × | × | × |
| iRS X X X X X X sce Last Visit" form) X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | | | | | | | | | |
| 2.20 X X X X X X X X X X X X Ense SAGE-324* X X X X X X X X X X X X X X X X X X X | C-SSRS<br>("Since Last Visit" form) | × | X | х | x | x | х | x | x |
| 2.20 X X X X X X X X X X X X X X X X X X X | | | | | | | | | |
| X X X X | ESS | X | X | X | X | x | X | x | X |
| X X X X | PWC-20 | | | | | | | x | X |
| | Dispense SAGE-3248 | x | X | X | X | X | X | | |

Sage Therapeutics, Inc. CONFIDENTIAL

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023)

| Assessment | | | Treatme | Treatment Period | | | Follow-u | Follow-up Period |
|---|---|---|---|---|---|---|---|---|
| Study Month | Month 9 | Month 12 | Month 15 | Mouth 18 | Month 21 | Month 24 to<br>Month 60<br>(Every<br>3 Months) | | EOT EOS<br>$3 (\pm 3)$ days $14 (\pm 3)$ days<br>after last dose after last dose<br>of SAGE-324 of SAGE-324 |
| Window (Weeks) | +2 | +2 | +2 | +2 | +2 | ±2 | | |
| SAGE-324 accountability | X | X | Х | X | x | X | X | Х |
| SAGE-324 administration b | | 4 | Administered once daily before bed | e daily before be | pe | | | |
| AEs/SAEs | | | | | X | | | |
| Concomitant medication | | | | | X | | | |

Abbreviations: AE = adverse event; C-SSRS = Columbia-Suicide Severity Rating Scale; ECG = electrocardiogram; EOS = End of Study; EOT = End of Freatment: IP = investigational product; MSE = mental state examination;

PWC-20 = 20-item Physician Withdrawal Checklist; SAE = serious adverse event; WOCBP = women of childbearing potential.

ECG, blood sample collection for Note: The suggested order of assessments during clinic visits is vital signs, assessments, and questionnaires.

clinical laboratory

<sup>a</sup> Complete physical examination and a comprehensive neurological examination, including MSEs, should be performed as clinically necessary (see Section 12.1.3). Targeted physical and neurological examinations should be performed as indicated by AEs.

D Weight assessed annually.

<sup>°</sup> Vital signs comprise heart rate, respiratory rate, temperature, and blood pressure. Systolic and diastolic blood pressure are to be measured after the participant has been supine for at least 5 minutes prior to the measurement. Orthostatic blood pressure and heart rate will also be measured after the participant has been in the supine position for at least 5 minutes and then repeated approximately 1 and 3 minutes after standing.

d ECGs will be collected and read locally. All ECGs must be performed after the participant has been in a supine position for at least 5 minutes

<sup>(</sup>biochemistry) at Screening and at additional timepoints at the discretion of the investigator. A serum sample for blood alcohol level will be collected at Chemistry, hematology, coagulation, and urinalysis at Screening and at all additional timepoints. Myoglobin (urinalysis) and serum creatine kinase Screening and all additional timepoints. HbA1c will be collected at every other scheduled visit.

<sup>&</sup>lt;sup>8</sup> If a participant experiences AEs at any time during the Treatment Period that are considered by the investigator to be related to the IP and not tolerable, the investigator may reduce the dose of IP in 15 mg decrements. Self-administration of IP will be interrupted for 3 to 8 days before the initiation of the reduced

b Participants will self-administer on an outpatient basis a single dose of SAGE-324 once daily in the evening before bed, with a snack if bedtime is not within 2 hours of the evening meal.

Statistical Analysis Plan Methods Version 1.0 22Oct2024 Protocol Number: 324-ETD-303 (Version 4.0 02 Nov 2023)

44

Sage Therapeutics, Inc. CONFIDENTIAL

# APPENDIX B. HANDLING OF MISSING DATES

Partial dates will adhere to the following conventions in order to classify TEAEs and to classify prior and concomitant medications.

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in derivation.

### Adverse Events

In the event of a missing/incomplete start or stop date associated with an adverse event, only the treatment-emergence will be imputed using the algorithm below. Dates will not be imputed.

In general, if the missing/incomplete start date is not clearly prior to initiation of treatment, then the AE will be considered a TEAE.

If the AE end date is prior to the initiation of treatment, the AE will not be considered a TEAE.

If the AE end date is on or after the initiation of treatment:

- If the AE start date is completely missing or if the year is missing, then the AE will be considered a TEAE
- For partial AE start dates:
  - Known year, unknown month and day (or known year and day, unknown month)
    - If the year is the same as or later than the year of the first dose, the AE will be considered a TEAE
    - Otherwise, the AE will not be considered a TEAE
  - Known year and month, unknown day
    - If the month and year are the same as or later than the month and year of the first dose, the AE will be considered a TEAE
    - Otherwise, the AE will not be considerd a TEAE

## Prior and Concomitant Medications

No imputation process will be used to estimate missing data, except for the purposes of classifying medications as prior and/or concomitant. The following algorithms will be used for partially missing dates.

For start dates of medication uses:

 The day and month are missing: if the participant started receiving the study dosing in the reported year, the first dosing date will be used as the start date; otherwise '01 January' will be used as the start date.

Sage Therapeutics, Inc. CONFIDENTIAL

The day is missing: if the participant started receiving the study dosing in the reported
month and year, the first dosing date will be used as the start date; otherwise, the first
day of the reported month and year will be used as the start date.

For stop dates of events or medication uses:

- The day and month are missing: if the study end date is in the reported year, the study
  end date will be used as the stop date; otherwise, '31 December' will be used as the
  stop date.
- The day is missing: if the study end date is in the reported month and year, the study
  end date will be used as the stop date; otherwise, the end of the reported month and
  year will be used as the stop date.

If a medication has the stop date completely missing or missing the year, this medication will be considered as ongoing and concomitant. If a participant is missing a treatment start date, medication will not be classified as either prior or concomitant.

Sage Therapeutics, Inc. CONFIDENTIAL

# APPENDIX C. LIST OF DISPLAYS

| Display Number | Display Title | Analysis Set Used |
|---|---|---|
| Tables | | |
| 14.1.1 | Disposition of Participants | All Participants |
| 14.1.2 | Analysis Sets | All Participants |
| 14.1.3.1 | Major Protocol Deviations | Safety Set |
| 14.1.3.2 | Protocol Deviations Related to COVID-19 | Safety Set |
| 14.1.4.1 | Demographics and Baseline Characteristics | Safety Set |
| 14.1.4.2 | Demographics and Baseline Characteristics - Subgroups | Safety Set |
| 14.1.5 | Summary of Disease History | Safety Set |
| 14.1.6 | Medical/Surgical History | Safety Set |
| 14.1.7.1 | Prior Medications | Safety Set |
| 14.1.7.2 | Concomitant Medications | Safety Set |
| 14.1.8.1 | Investigational Product Exposure | Safety Set |
| 14.1.8.2 | Total Exposure Duration by Dose at<br>Investigational Product Discontinuation | Safety Set |
| 14.1.8.3 | Investigational Product Adherence | Safety Set |

| 14.3.1.1 | Summary of Treatment-Emergent Adverse<br>Events | Safety Set |
|---|---|---|
| 14.3.1.2 | Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety Set |
| 14.3.1.3 | Treatment-Emergent Adverse Events by<br>Preferred Term | Safety Set |

| 14.3.1.4 Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Set 14.3.1.5 Treatment-Emergent Adverse Events Leading to Investigational Product Discontinuation by System Organ Class and Preferred Term Safety Set 14.3.1.6 Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term Safety Set 14.3.1.7 Treatment-Emergent Adverse Events by Maximum Severity Safety Set 14.3.1.8 Treatment-Emergent Adverse Events by Maximum Relationship to Investigational Product Safety Set 14.3.1.9 Serious Treatment-Emergent Adverse Events by Preferred Term Safety Set 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests Safety Set 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline Safety Set 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.3.1 Summary o | | | |
|---|---|---|---|
| Leading to Investigational Product Discontinuation by System Organ Class and Preferred Term 14.3.1.6 Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term 14.3.1.7 Treatment-Emergent Adverse Events by Maximum Severity 14.3.1.8 Treatment-Emergent Adverse Events by Maximum Relationship to Investigational Product 14.3.1.9 Serious Treatment-Emergent Adverse Events by Preferred Term 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.1.4 | Events by System Organ Class and | Safety Set |
| Leading to Study Discontinuation by System Organ Class and Preferred Term 14.3.1.7 Treatment-Emergent Adverse Events by Maximum Severity 14.3.1.8 Treatment-Emergent Adverse Events by Maximum Relationship to Investigational Product 14.3.1.9 Serious Treatment-Emergent Adverse Events by Preferred Term 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.1.5 | Leading to Investigational Product Discontinuation by System Organ Class | Safety Set |
| Maximum Severity 14.3.1.8 Treatment-Emergent Adverse Events by Maximum Relationship to Investigational Product 14.3.1.9 Serious Treatment-Emergent Adverse Events by Preferred Term Summary of Clinical Chemistry Safety Set 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.2.3 Safety Set | 14.3.1.6 | Leading to Study Discontinuation by | Safety Set |
| Maximum Relationship to Investigational Product 14.3.1.9 Serious Treatment-Emergent Adverse Events by Preferred Term 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.1.7 | | Safety Set |
| Events by Preferred Term 14.3.4.1.1 Summary of Clinical Chemistry Safety Set 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.1.8 | Maximum Relationship to Investigational | Safety Set |
| 14.3.4.1.2 Shift of Clinical Chemistry Safety Set 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.2.3 Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.1.9 | | Safety Set |
| 14.3.4.1.3 Potentially Clinically Significant (PCS) Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.1.1 | Summary of Clinical Chemistry | Safety Set |
| Values in Clinical Chemistry Excluding Liver Function Tests 14.3.4.1.4 Potentially Clinically Significant (PCS) Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Values in Hematology 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.1.2 | Shift of Clinical Chemistry | Safety Set |
| Values in Liver Function Tests Any Time Post-baseline 14.3.4.2.1 Summary of Hematology Safety Set 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Safety Set Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.1.3 | Values in Clinical Chemistry Excluding | Safety Set |
| 14.3.4.2.2 Shift of Hematology Safety Set 14.3.4.2.3 Potentially Clinically Significant (PCS) Safety Set Values in Hematology Safety Set 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.1.4 | Values in Liver Function Tests Any Time | Safety Set |
| 14.3.4.2.3 Potentially Clinically Significant (PCS) Safety Set Values in Hematology 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.2.1 | Summary of Hematology | Safety Set |
| Values in Hematology 14.3.4.3.1 Summary of Coagulation Safety Set | 14.3.4.2.2 | Shift of Hematology | Safety Set |
| | 14.3.4.2.3 | | Safety Set |
| 14.3.4.3.2 Shift of Coagulation Safety Set | 14.3.4.3.1 | Summary of Coagulation | Safety Set |
| | 14.3.4.3.2 | Shift of Coagulation | Safety Set |

| 14.3.4.3.3 | Potentially Clinically Significant (PCS)<br>Values in Coagulation | Safety Set |
|---|---|---|
| 14.3.4.4.1.1 | Summary of Urinalysis, Continuous<br>Parameters | Safety Set |
| 14.3.4.4.1.2 | Summary of Urinalysis, Categorical<br>Parameters | Safety Set |
| 14.3.4.4.2 | Shift of Urinalysis | Safety Set |
| 14.3.4.5.1 | Summary of 12-Lead Electrocardiogram | Safety Set |
| 14.3.4.5.2 | Shift of Overall Electrocardiogram<br>Interpretation | Safety Set |
| 14.3.4.5.3 | Potentially Clinically Significant (PCS)<br>QTcF Values | Safety Set |
| 14.3.4.6.1 | Summary of Vital Signs | Safety Set |
| 14.3.4.6.2 | Potentially Clinically Significant (PCS)<br>Values in Vital Signs | Safety Set |
| 14.3.4.7.1 | Summary of Columbia-Suicide Severity<br>Rating Scale | Safety Set |
| 14.3.4.7.2 | Shift From Baseline in Columbia-Suicide<br>Severity Rating Scale (C-SSRS) Suicidal<br>Ideation and Suicidal Behavior by Study<br>Visit | Safety Set |
| 14.3.4.7.3 | Shift From Baseline in Columbia-Suicide<br>Severity Rating Scale (C-SSRS) Maximum<br>Severity Score in Suicidal Ideation at Any<br>Time Post-baseline | Safety Set |
| 14.3.4.8 | Summary of Physician Withdrawal<br>Checklist (PWC-20) | Safety Set |
| 14.3.4.9.1 | Summary of Epworth Sleepiness Scale –<br>Individual Items | Safety Set |
| 14.3.4.9.2 | Summary of Epworth Sleepiness Scale –<br>Total Score | Safety Set |

| Listings | | |
|---|---|---|
| 16.2.1.1 | Participant Disposition | All Participants |
| 16.2.1.2 | Screen Failures | Screen Failure<br>Participants |
| 16.2.2.1 | Inclusion/Exclusion Criteria Violations | All Participants,<br>Excluding Screen<br>Failures |
| 16.2.2.2 | Protocol Deviations | Safety Set |
| 16.2.3 | Analysis Sets | All Participants |
| 16.2.4.1 | Demographics and Informed Consent | Safety Set |
| 16.2.4.2 | Child-bearing Potential | Safety Set |
| 16.2.4.3.1 | Medical/Surgical History | Safety Set |
| 16.2.4.3.2 | Essential Tremor Disease History | Safety Set |
| 16.2.4.4.1 | Prior Medications | Safety Set |
| 16.2.4.4.2 | Concomitant Medications | Safety Set |
| 16.2.4.5 | Concomitant Procedures | Safety Set |
| 16.2.5.1 | Investigational Product Dispensation and<br>Return | Safety Set |
| 16.2.5.2.1 | Investigational Product Administration –<br>Daily Dosing Diary | Safety Set |
| 16.2.5.2.2 | Investigational Product Administration –<br>Log Records | Safety Set |
| 16.2.5.3 | Investigational Product Exposure and<br>Adherence | Safety Set |



| 16.2.8.2.5 | Central Laboratory Drug Screen | Safety Set |
|------------|----------------------------------------------------|------------|
| 16.2.8.3 | 12-Lead Electrocardiogram (ECG) | Safety Set |
| 16.2.8.4 | Vital Signs | Safety Set |
| 16.2.8.5 | Physical Examinations | Safety Set |
| 16.2.8.6 | Mental Status Examination | Safety Set |
| 16.2.8.7 | Abbreviated Neurological Examination | Safety Set |
| 16.2.8.10 | Columbia-Suicide Severity Rating Scale<br>(C-SSRS) | Safety Set |
| 16.2.8.11 | Physician Withdrawal Checklist | Safety Set |
| 16.2.8.12 | Epworth Sleepiness Scale | Safety Set |

# Certificate Of Completion

Envelope Id: 1171D0B2DF2443FCAB7EBD0FEEFD3DF8

Subject: Sage\_324-ETD-303\_sap\_v1.0\_20241022\_methods.pdf

Source Envelope:

Document Pages: 53 Certificate Pages: 6

Signatures: 7 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator:

IP Address:

## Record Tracking

Status: Original

23-Oct-2024 | 09:29

Holder:

Location: DocuSign

Sent: 23-Oct-2024 | 09:32 Resent: 23-Oct-2024 | 20:53 Viewed: 24-Oct-2024 | 08:44 Signed: 24-Oct-2024 | 08:45

Timestamp

# Signer Events

Sage Therapeutics

Security Level: Email, Account Authentication

(Required)

# Signature



Signature Adoption: Uploaded Signature Image

Signature ID:

28381C0A-811F-448C-A297-569013A4FF00

With Signing Authentication via DocuSign password

# Electronic Record and Signature Disclosure:

Not Offered via DocuSign



Sage Therapeutics - Part 11

Security Level: Email, Account Authentication (Required)





Using IP Address:

With Signing Reasons (on each tab): I approve this document

> Sent: 23-Oct-2024 | 09:32 Viewed: 23-Oct-2024 | 11:22 Signed: 23-Oct-2024 | 11:23

Sent: 23-Oct-2024 | 09:32 Resent: 23-Oct-2024 | 20:53 Viewed: 23-Oct-2024 | 21:09

Signature Adoption: Pre-selected Style

Signature ID:

95A42B3B-78C2-4820-B3C9-63A26F4312B3

Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

# Electronic Record and Signature Disclosure:

Not Offered via DocuSign



Sage Therapeutics - Part 11

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

104D24A1-5373-4DB6-9066-E2ED46A7602E

Using IP Address:

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure:



Signer Events
Not Offered via DocuSign

Sent: 23-Oct-2024 | 09:32
Viewed: 23-Oct-2024 | 09:37
Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style
Signature ID:
4CB4D7BF-3097-4239-AC1B-C40A2362AF78
Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

Electronic Record and Signature Disclosure: Accepted: 20-Jul-2021 | 11:15 ID: fd75acbc-bffa-47ad-933d-bb55286e892e

Security Level: Email, Account Authentication (Required)

Sent: 23-Oct-2024 | 09:32 Viewed: 23-Oct-2024 | 09:36 Signed: 23-Oct-2024 | 09:37

Signature Adoption: Pre-selected Style
Signature ID:
B8851932-B1EB-4F32-B640-96A5FE300A64
Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

Electronic Record and Signature Disclosure: Not Offered via DocuSign



Security Level: Email, Account Authentication (Required)



Sent: 23-Oct-2024 | 09:32 Viewed: 23-Oct-2024 | 09:53 Signed: 23-Oct-2024 | 11:50

Signature Adoption: Pre-selected Style
Signature ID:
67C05255-8C9B-4377-9514-2BB8E4ABBAE9
Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

Electronic Record and Signature Disclosure: Not Offered via DocuSign





Sent: 23-Oct-2024 | 09:32 Viewed: 23-Oct-2024 | 09:52 Signed: 23-Oct-2024 | 09:54

Signature Adoption: Pre-selected Style
Signature ID:
3EEED344-DA9D-425B-9915-C78423F5271E
Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

| Signer Events | Signature | Timestamp |
|---|---|---|
| Electronic Record and Signature Disclosure:<br>Not Offered via DocuSign | | |
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 23-Oct-2024 09:32 |
| Certified Delivered | Security Checked | 23-Oct-2024 09:52 |
| Signing Complete | Security Checked | 23-Oct-2024 09:54 |
| Completed | Security Checked | 24-Oct-2024 08:45 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disc | losure | |

## ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Sage Therapeutics - Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

# All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# How to contact Sage Therapeutics - Part 11:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to:

# To advise Sage Therapeutics - Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from Sage Therapeutics - Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with Sage Therapeutics - Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

 decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Sage Therapeutics Part 11 as described above, you consent to
  receive exclusively through electronic means all notices, disclosures, authorizations,
  acknowledgements, and other documents that are required to be provided or made
  available to you by Sage Therapeutics Part 11 during the course of your relationship
  with Sage Therapeutics Part 11.